CLINICAL TRIAL: NCT05317182
Title: "Comparative Study of the Accuracy of Dental Contacts of an Occlusal Splint Made According to Conventional or Digital Techniques Using GeoMagic®."
Brief Title: Accuracy of Dental Contacts of an Occlusal Splint Made According to Conventional or Digital Techniques Using GeoMagic®.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Alvaro Blasi, Principal investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Other
Other Study IDs: REST-ECL-2021-07
Record Dates: First submitted 2022-03-06; First posted 2022-04-07 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Occlusal Splints
Keywords: Digital Dentistry; Occlusal records; Intraoral scan

STUDY DESIGN:
Intervention Model Description: This clinical study has three arms of equal size: occlusal splints made by conventional impression and conventional fabrication (Group 1), occlusal splints made by conventional impression and digital design and fabrication (Group 2), and occlusal splints performed by intra-oral scanner and digital design and fabrication (Group 3).
  Otherwise, the allocation of each subject to each group will be done at random by a list made with specialized software until the sample will be fulfilled when the patient is recruited.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Analogic-Analogic (Active Comparator): Occlusal splints made by conventional impression and conventional fabrication.
  Interventions: Other: Occlusal Splints Analogic-Analogic
- Analogic-Digital (Active Comparator): Occlusal splints made by conventional impression and digital design and fabrication.
  Interventions: Other: Occlusal Splints Analogic-Digital
- Digital-Digital (Active Comparator): Occlusal splints performed by intra-oral scanner and digital design and fabrication.
  Interventions: Other: Occlusal Splints Digital-Digital

INTERVENTIONS:
Other: Occlusal Splints Analogic-Analogic — Take a conventional impression to the patient and conventional fabrication of the splint.
  Arms: Analogic-Analogic
Other: Occlusal Splints Analogic-Digital — Take a conventional impression to the patient and digital fabrication of the splint.
  Arms: Analogic-Digital
Other: Occlusal Splints Digital-Digital — Take a digital impression to the patient and digital fabrication of the splint.
  Arms: Digital-Digital

SUMMARY:
To compare the accuracy of the occlusal splints made by conventional impression and milled with the splint made by intraoral scanner and milled.

DETAILED DESCRIPTION:
Forty participants received two different occlusal devices from two different workflows (fully conventional and fully digital). Every splint was scanned before and after the occlusal adjustments in order to compare the volumetric changes. Furthermore, the scans were compared in a software Geomagic® Control X calculates and measures the distance from every surface point from the initial dataset (occlusal devices before adjustment) to the final dataset (occlusal device after adjustment).

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 to 70 years old.
* Patients who maintain until first molar in both arches.
* Patients who need occlusal splints due to bruxism.

Exclusion Criteria:

* Pregnant patients.
* Patients with removable prostheses.
* Patients with fixed prostheses between six to six in both arches.
* Patients with partial edentulism, do not maintain until first molar in both arches.
* Patients with Temporomandibular Disorders (TMD): articular noises, pain on palpation, limited opening.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Volumetric changes assessed in Root Mean Square (RMS) | 1 week
  The software of automatically graphical comparisons called Geomagic® Control X (Geomagic Inc., 3D Systems Inc., USA) will be used to calculate the accuracy by measuring the distance (positive or negative) from every surface point from the initial dataset (occlusal devices before adjustment) to the final dataset (occlusal device after adjustment). This approach will give us the mean of the simple arithmetic difference.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Roig, DDS, PhD, Study Director — Universitat Internacional de Catalunya
Locations (1):
- Blasi Clinica Dental Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Blasi A, Henarejos-Domingo V, Palacios-Banuelos R, Aparicio C, Roig M. Comparison accuracy of digital and analog method using milled occlusal splints. J Esthet Restor Dent. 2023 Oct;35(7):1103-1112. doi: 10.1111/jerd.13039. Epub 2023 Mar 21. PMID 36942721